CLINICAL TRIAL: NCT01586572
Title: Comparison of Immunogenicity of Type 1 mOPV Administered at Short Intervals With Type 1 mOPV1 and Type 1 & 3 bOPV Oral Polio Vaccine Given at Standard Intervals in Pakistan:A Randomized Trial
Brief Title: Pakistan Short Interval mOPV1 Compared With Standard Interval mOPV1 and bOPV 1,3
Acronym: SIAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Anita Kaniz Mehdi Zaidi, Professor and Chairperson, Pediatrics and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1891-Ped-ERC-11
Record Dates: First submitted 2012-04-02; First posted 2012-04-27 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Polio
Keywords: Polio virus type 1,2,3; Poliovaccine-Oral; Poliovaccine; Trivalent Oral Polio vaccine; Monovalent oral polio vaccine; Bivalent Oral polio vaccine
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- mOPV1- Arm A (Experimental): Arm A will be administered a second dose of mOPV1 seven days after the 42 day mOPV1 index dose.Second dose of tOPV2 will be given at day 79.
  Interventions: Drug: mOPV1
- mOPV1- Arm B (Experimental): Arm B will be administered a second dose of mOPV1 fourteen days after after the 42 day mOPV1 index dose.Second dose of tOPV2 will be given at 86 days.
  Interventions: Drug: mOPV1
- mOPV1-Arm C (Experimental): Arm C will receive the second dose of mOPV1 thirty days after the 42 day mOPV1 index dose.Second dose of tOPV2 will be given at 102 days.
  Interventions: Drug: mOPV1
- Arm D- bOPV1,3 (Experimental): Arm D will be administered a second dose of bOPV1,3 thirty days after the 42 day bOPV1,3 index dose.Second dose of tOPV2 will be given at day 102.
  Interventions: Drug: bOPV 1,3

INTERVENTIONS:
Drug: mOPV1 — Monovalent type 1 oral poliovirus vaccine (mOPV1) containing at least106 TCID50 of Sabin- strain poliovirus type 1.
  Other Names: Monovalent type 1 oral poliovirus vaccine
  Arms: mOPV1- Arm A; mOPV1- Arm B; mOPV1-Arm C
Drug: bOPV 1,3 — The bivalent vaccine containing at least 106 CCID50 of Sabin poliovirus type 1 and 105•8 CCID50 of Sabin poliovirus type 3.
  Other Names: Bivalent Oral Polio Vaccine
  Arms: Arm D- bOPV1,3

SUMMARY:
Globally, polio cases have decreased by over 99% since 1988. However, wild poliovirus cases continue in Pakistan. Conflict and lack of access to children due to on-going insecurity in tribal areas present special challenges in interrupting transmission rapidly. There exists limited knowledge on the effect of shorter intervals of mOPV vaccination on immunogenicity levels in young children. The aim of this study is to demonstrate the non-inferiority of shorter intervals (7 and 14 days) between doses of mOPV1 vaccine compared to the customary interval (30 days). A 4th arm will receive bivalent (bOPV) vaccine at standard intervals beginning at 6 weeks of age.

DETAILED DESCRIPTION:
This randomized clinical trial which will be conducted in 5 low-income areas in and around Karachi (4 peri-urban, contiguous coastal villages outside Karachi, and one urban squatter settlement) where the Aga Khan University's Department of Paediatrics and Child Health has well-established demographic surveillance with all pregnancies and new births in the area captured through the system. The study participants will be enrolled from birth until 102 days. Subjects will be randomized to one of four trial arms.

All children will receive tOPV at birth. At 42 days (6 weeks) of age, three study arms will receive a dose of mOPV1 whereas the fourth arm will receive a dose of bOPV1&3 as per protocol. Then 7 or 14 or 30 days later, the study participants in Arms A, B, and C will receive a second dose of mOPV1 while a second dose of bOPV 1&3 will be given to participants in Arm D at 30 days.

Name and description of products:

1. Standard trivalent oral poliovirus vaccine (tOPV), in a 10:1:6 formulation, containing at least 106 TCID50 of Sabin -strain poliovirus type 1, at least 105 TCID50 of Sabin-strain poliovirus type 2 and at least 105.8 TCID50 of Sabin-strain poliovirus type 3.
2. Monovalent type 1 oral poliovirus vaccine (mOPV1) containing at least106 TCID50 of Sabin- strain poliovirus type 1.
3. The bivalent oral polio vaccine containing at least 106 CCID50 of Sabin poliovirus type 1 and 105•8 CCID50 of Sabin poliovirus type 3.

Sample Size:

To show non-inferiority of a 2-dose mOPV1 schedule with shorter-intervals (either 7 or 14 days) [intervention] compared to a 2-dose mOPV1 schedule administered at 30-day intervals [control], and a 2-dose bOPV13 schedule administered at a 30-day interval (control) assuming a power of 0.90 (beta) and p of 0.05 (alpha), we require a sample of 139 for each study group, for a total of 556 subjects. To compensate for drop out, attrition and insufficient sera for laboratory testing, an inflated (by ~ 50%) sample size of 200 in each group will be used (total sample size of 800)

Efficacy Endpoints:

The primary endpoint is seroconversion with antibodies to poliovirus type 1 following a two-dose schedule of mOPV1 given at intervals of 7 and 14 days compared to mOPV1 and bOPV1&3 given at the standard interval of 30 days..

The secondary endpoint is seroconversion following the birth dose of tOPV.

All samples will be processed at the Centers of Disease Control and Prevention CDC) Laboratories (a Global Specialized Polio Network Laboratory).

ELIGIBILITY:
Inclusion Criteria:

* Infants > 2.5 kg birth weight
* Immediate cry
* No neonatal IMCI danger signs
* Not planning to travel away during entire the study period (birth-102 days)

Exclusion Criteria:

* High-risk newborns will be excluded, as well as newborns requiring hospitalization
* Birth weight below 2.5 kg
* Cry >2 minutes
* With any neonatal IMNCI danger signs
* Residence >30 km from study site
* Family is planning to be absent during the birth - 102 day study period.
* A diagnosis or suspicion of immunodeficiency disorder (either in the participant or in a member of the immediate family - e.g. several early infant deaths, household member on chemotherapy) will render the newborn ineligible for the study.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2012-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Seroconversion with antibodies to poliovirus type 1 following a two-dose schedule of mOPV1 given at intervals of 7 and 14 days compared to mOPV1 and bOPV1&3 given at the standard interval of 30 days. | Participants will be followed till 102 days after birth
  Humoral immunity: Sera collected at birth (cord blood or peripheral blood), at 42 days, at 79 days, at 86 days, or at 102 days (depending on study arm) will be examined for the presence (detectable) or absence of neutralizing antibodies to all three poliovirus serotypes. A reciprocal titer of >8 is considered to indicate the presence of neutralizing antibodies. For participants with detectable antibodies, seroconversion is defined as a 4-fold increase over the expected decline of maternally-derived antibodies (half-life assumed to be 28 days).

SECONDARY OUTCOMES:
Seroconversion following the birth dose of tOPV. | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Anita KM Zaidi, MD; MSc, Principal Investigator — Aga Khan University; Fatima FM Mir, MBBS, Study Director — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Mir F, Quadri F, Mach O, Ahmed I, Bhatti Z, Khan A, Rehman NU, Durry E, Salama M, Oberste SM, Weldon WC, Sutter RW, Zaidi AK. Monovalent type-1 oral poliovirus vaccine given at short intervals in Pakistan: a randomised controlled, four-arm, open-label, non-inferiority trial. Lancet Infect Dis. 2015 Aug;15(8):889-97. doi: 10.1016/S1473-3099(15)00093-6. Epub 2015 Jun 17. PMID 26093979